CLINICAL TRIAL: NCT01494766
Title: Pilot Study of the Efficacy of Tyrosine in Restless Legs Syndrome
Brief Title: Efficacy of Tyrosine in Restless Legs Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-11-146
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Restless Legs Syndrome (RLS)
Keywords: RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Tyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tyrosine (Other): Dietary Supplement: L-Tyrosine
  Other Names:
  NOW Brand L-Tyrosine 750 mg Tablets
  -Tyrosine 750 mg PO every day for 7 days, then increase to 1500 mg PO every day for 7 days, then increase to 2250 mg PO every day for 7 days, then increase to 3000 mg PO every day for remainder of the study.
  Interventions: Dietary Supplement: L-Tyrosine

INTERVENTIONS:
Dietary Supplement: L-Tyrosine — L-Tyrosine 750 mg PO every day for 7 days, then increase to 1500 mg PO every day for 7 days, then increase to 2250 mg PO every day for 7 days, then increase to 3000 mg PO every day for remainder of the study.
  Other Names: NOW Brand L-Tyrosine 750 mg Tablets

SUMMARY:
Tyrosine is a non essential amino acid that is the precursor of the neurotransmitter, dopamine. Tyrosine is converted into Levodihydrophenylalanine (L-Dopa) and L-Dopa is subsequently and avidly converted into dopamine. It is well known that dopamine deficiency leads to the manifestations of restless legs syndrome (RLS). Studies have shown dopamine agonists and L-dopa to be effective in controlling symptoms. No studies to date have been done to determine the role of tyrosine in RLS. This open-label pilot study aims to determine the efficacy and tolerability of tyrosine in RLS, as current agents have limitations in treating RLS in addition to adding another possible agent to the investigators arsenal of treating RLS that maybe more cost efficient. In this pilot study, the dose of tyrosine will be escalated from 750 mg once daily by mouth (PO) up to 3000 mg once daily PO, as tolerated, in increments of 750 mg every week in patients who meet the inclusion criteria for RLS. Patients' symptoms will be monitored on a weekly basis for six weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 80 years and
2. Newly diagnosed (medication-naïve) as having restless legs syndrome (using the International Restless Legs Syndrome Study Group (IRLSSG20) diagnostic criteria with a score of greater than or equal to 15, see Appendix A) and
3. That interfered with sleep onset and/or maintenance for greater than four nights/week for a minimum of six months
4. Currently not receiving treatment for RLS

Exclusion Criteria:

1. Patients suffering from secondary RLS (other movement and/or primary sleep disorders, chronic renal insufficiency - calculated from the creatinine clearance, and/or iron deficiency - baseline serum ferritin level less than 10 ng/ml)
2. Patients currently on pharmacotherapy for RLS (not medication-naïve) or previous use of pharmacotherapy for RLS in the past
3. Patients that are pregnant and/or breastfeeding
4. Patients that are on levothyroxine or monoamine oxidase inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
International RLS Survey Group (IRLSSG20) Score | 6 weeks
  Use of this survey to be used as a marker for severity of RLS symptoms and therefore efficacy of this medication.

SECONDARY OUTCOMES:
Clinical global impression-global improvement (CGI-I) scale | 6 weeks
  Use of the CGI-I scale as a secondary outcome measure to determine severity of RLS symptoms and efficacy of medication.
Medical Outcomes Study - Sleep Scale (MOS-SS) | 6 weeks
  Use of the MOS-SS to determine severity of RLS symptoms and efficacy of medication.
Case Report Form | 6 weeks
  Use of a history and physical examination (limited neurological exam) to be used as a secondary assessment measure of RLS symptom severity and medication efficacy. They will be charted in case report format.

CONTACTS AND LOCATIONS:
Locations (1):
- Seton Family of Hospitals, Austin, Texas, United States